CLINICAL TRIAL: NCT00185848
Title: Imaging the Biodistribution of the Positron Emission Tomography Reporter Probe, [18F]FHBG, in Humans.
Brief Title: Assessing the Suitability of an Imaging Probe for Use in Clinical Cell and Gene Therapy Trials in Cancer and Rheumatoid Arthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanjiv Sam Gambhir (Other)
Responsible Party: Sponsor-Investigator, Sanjiv Sam Gambhir, Virginia and D.K. Ludwig Professor for Clinical Investigation in Cancer Research, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BRNCNS0003; 95908 (Other: Stanford University Alternate IRB Approval Number); BRNCNS0003 (Other: Stanford University)
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Brain Cancer; Arthritis, Rheumatoid; Central Nervous System Neoplasms; Glioma
MeSH Terms: conditions — Brain Neoplasms; Arthritis, Rheumatoid; Central Nervous System Neoplasms; Glioma | interventions — 9-(4-fluoro-3-hydroxymethylbutyl)guanine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- [18F]FHBG arm (Experimental)
  Interventions: Radiation: [18F]FHBG

INTERVENTIONS:
Radiation: [18F]FHBG — < 7mCi and 2 ug, iv
  Other Names: 18F-FHBG

SUMMARY:
The purpose of this study is to determine whether [18F]FHBG is suitable for use as an imaging probe in cancer or rheumatoid arthritis patients enrolled in cell or gene therapy trials. In this phase 1 study we will assess the safety and biodistribution of [18F]FHBG in patients.

DETAILED DESCRIPTION:
The success of cell and gene therapy depends on specific targeting of the therapeutic gene or cell that is administered to the patient. Our goal is to develop an imaging method to non-invasively monitor the location of the therapeutic gene or cell. Imaging should help in the design of better protocols and potentially reduce side-effects of cell and gene therapy.

ELIGIBILITY:
Inclusion Criteria:

- Clinical diagnosis of brain tumor or rheumatoid arthritis

Exclusion Criteria:

- Below 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2005-04; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of the study for each patient is acquisition of PET/CT image. | Time of scan

SECONDARY OUTCOMES:
Collection of vital signs, EKG, blood chemistry and CBC data | day 1, 2 and 8.

CONTACTS AND LOCATIONS:
Overall Officials: Sanjiv Sam Gambhir M.D., Ph.D., Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - University of California Los Angeles, Los Angeles, California
  - Stanford University School of Medicine, Stanford, California

REFERENCES:
- [Background] Yaghoubi S, Barrio JR, Dahlbom M, Iyer M, Namavari M, Satyamurthy N, Goldman R, Herschman HR, Phelps ME, Gambhir SS. Human pharmacokinetic and dosimetry studies of [(18)F]FHBG: a reporter probe for imaging herpes simplex virus type-1 thymidine kinase reporter gene expression. J Nucl Med. 2001 Aug;42(8):1225-34. PMID 11483684